CLINICAL TRIAL: NCT04513834
Title: Efficacy of a Multi-faceted Intervention Combining an Educational Outreach Visit to General Practitioners and Patient Education Material to Deprescribe Proton Pump Inhibitors (PPI): a Population-based, Pragmatic, Cluster-randomized Controlled Trial
Acronym: DeprescrIPPDAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: RC20_0339
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Proton Pump Inhibitors; Deprescription
Keywords: Proton pump inhibitors; Deprescription; Multi-faceted intervention; Patient-centered; Primary health care; Pharmacoepidemiology

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multi-faceted intervention (Experimental): Patient education material on PPI deprescribing will be sent to the patients and their general practitioner (GP) will receive an educational outreach visit by a Delegue d'Assurance Maladie (DAM, healthcare representative )
  Interventions: Other: GP will receive the educational outreach visit by a DAM (healthcare representative).; Other: Patient education material on PPI deprescribing will be sent to the patients
- Educational outreach visit to GPs (Active Comparator): GP will receive the educational outreach visit by a DAM (healthcare representative). Their patients will not receive any patient education material.
  Interventions: Other: GP will receive the educational outreach visit by a DAM (healthcare representative).
- Control (No Intervention): Neither the patients nor their GP will receive any information.

INTERVENTIONS:
Other: GP will receive the educational outreach visit by a DAM (healthcare representative). — GP will receive the educational outreach visit by a DAM (healthcare representative).
  Arms: Educational outreach visit to GPs; Multi-faceted intervention
Other: Patient education material on PPI deprescribing will be sent to the patients — Patient education material on PPI deprescribing will be sent to the patients
  Arms: Multi-faceted intervention

SUMMARY:
Deprescribing is defined as "the process of withdrawal of an inappropriate medication, supervised by a health care professional with the goal of managing the polypharmacy and improving outcomes". Inappropriate use of proton pump inhibitors (PPI) is associated with severe adverse drug reactions and a major economic impact. Deprescribing should be considered when inappropriate prescription of PPI is identified.

DeprescrIPP DAM is a pragmatic trial, population-based, designed in clusters. It wil assess the efficacy of a multi-faceted intervention (an educational outreach visit to general practitioners associated with the sending of patient education material to their patients) to deprescribe PPI.

ELIGIBILITY:
Inclusion Criteria:

* General practitioners (GP)

  • All GP settled in the French region Pays-de-la-Loire having seen more than 100 different patients in the year before baseline, will be eligible.
* Patients

  * Aged more than 18 years old
  * Affiliated to the French health insurance CPAM
  * Treated with PPI> 300DDD/year in the year before baseline (estimated with reimbursement databases).
  * Whose GP is included in the study

Exclusion Criteria:

* General practitioners (GPs) :

  • Participation refusal
* Patients

  * Participation refusal
  * Patients at risk of gastroduodenal lesions i.e. treated with nonsteroidal anti-inflammatory drugs (NSAIDs) and over 65 years old or treated with either corticosteroids or anticoagulants or platelet aggregation inhibitors
  * Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25000 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
PPI deprescribing | 12 months
  Proportion of patients achieving a 50% decrease in their reimbursement of PPI (Defined Daily Dose (DDD)/year) at the end of the intervention compared to baseline (estimated with reimbursement databases)

SECONDARY OUTCOMES:
Characteristics of patients engaging in the deprescription process | 12 months
  Sex, age, long-term illness, universal health insurance, complementary health insurance, medication

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No